CLINICAL TRIAL: NCT07247331
Title: Effect of Action Observation Therapy on Spasticity, Gross Motor Function, Balance And Participation in Children With Cerebral Palsy: A Randomized Controlled Study
Brief Title: The Effect of Action Observation Therapy on Spasticity, Motor Function, and Balance in Children With Cerebral Palsy
Acronym: AOT-CP
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Merve Yıldız, physiotherapist, Suleyman Demirel University
Other Study IDs: suleymanedu//Myildiz001
Record Dates: First submitted 2024-01-04; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Cerebral Palsy; Spastic Diplegia Cerebral Palsy; Hemiplegic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy; Cerebral palsy, spastic, diplegic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treatment Program of the Control Group (Group 1):: Treatment Program of the Control Group (Group 1): This group will not be shown any video clips, and general physiotherapy methods will be applied to their current needs, 2 sessions a week for 6 weeks. This method includes stretching exercises for spastic muscles, strengthening exercises for the antagonist of the spastic muscle, and stabilization exercises.
  Interventions: Other: action observation therapy
- Group 2: Action Observation Therapy for the lower extremities will be applied to this group by their parents at home, 2 sessions a week for 6 weeks. Participants will be shown a video of a task by their parents at home. The video to be watched will include a total of 6 activities planned to be watched every week. These 6 activities; squatting and getting up by picking up an object from the ground, walking 10 steps between parallel lines, transferring weight forward with the right and left feet, walking 5 steps sideways to the right and left, kicking the ball, climbing the step from the front and side. The video clips will be watched 3 times and after a 1-minute rest following each viewing, the participants will be asked to repeat each activity in the videos 3 times and at the end of each clip.
  Interventions: Other: action observation therapy
- Group 3: Children with spastic hemiparetic and diparetic CP included in our study were asked to watch and then perform the 6 activities in the video recording on a 10.2-inch tablet screen. The EGT program was applied for 20 minutes per day, 2 sessions per week for 6 weeks. Since there is no definitive protocol for children with diparetic CP, the EGT program applied is compatible with the protocol described by Sgandurra et al. In the application, the patient was asked to watch the activities in the video clip under the supervision of a physiotherapist, and after a one-minute rest period following each viewing, to repeat these activities physically actively for the duration of the video. After each EGT session, a 20-minute physiotherapy session was applied with a physiotherapist for the targets of the 6 activities. The scope of the applied physiotherapy consisted of activity-based exercises for the lower extremity, such as taking steps, weight transfer, balance and functionality.
  Interventions: Other: action observation therapy

INTERVENTIONS:
Other: action observation therapy — Action Observation Therapy (AOT) is among the neurorehabilitation approaches that enable motor learning by facilitating neuroplasticity. AOT is based on neuroscience and activation of the mirror neuron system. AOT occurs in the form of the observer following the motor action and performing the observed actions after observing the actions. AOT aims to improve different motor functions by providing motor learning through neuroplasticity activation.

SUMMARY:
In our randomized controlled study, which aims to investigate the contribution of Action Observation Therapy to rehabilitation by examining the effect of Action Observation Therapy on spasticity, gross motor function, balance and participation in children with spastic diplegic and hemiplegic cerebral palsy, the effectiveness of Action Observation Therapy to be applied in the home environment and accompanied by a physiotherapist will be investigated.

DETAILED DESCRIPTION:
In this study, G*Power 3.1.3 program was used to calculate the minimum sample size in each group (control group (group 1), group 2 and group 3), in other words, the number of individuals in the groups. In this context, the effect size was taken as d = 1.1, the significance level was α = 0.05, and the minimum number of individuals in each group was calculated as 11 (33 in total) for a power of 0.80 (80%). Similar studies (Sgandurra 2013, Kim 2018) were taken into consideration in obtaining these parameters. The number of individuals in each group (+10%) was planned to be at least 12 (36 in total), taking into account individuals who were missing, incorrect or excluded from the study.

In order to prevent bias in terms of participants meeting the inclusion criteria, sociodemographic and clinical characteristics, criteria such as age, cerebral palsy type, GMFCS level and presence of comorbidities were taken into account in assigning individuals to groups in the study, and the stratified randomization method will be used. Accordingly, the age ranges are taken as 5-7, 8-10, 11-13, and the cerebral palsy type is; spastic diplegic and hemiplegic, GMFCS level; It will be taken as I-III and the stratification process will be done accordingly. Before the study, written and verbal "Informed Consent Form" will be obtained from the parents of all participants in the study and control groups. The content of the study will be explained to the children who will participate in the study in a way that the child can understand, and the child's consent will be obtained. After recording the sociodemographic data of the participants for both the experimental and control groups, their spasticity was measured by the Modified Ashworth Scale (MAS), their gross motor function levels were measured by the Gross Motor Function Measurement (GMFM), their participation was measured by the Child and Adolescent Participation Survey (CASP), and their balance was measured by the Timed Up and Go Test ( TUG), Pediatric Reach Test (PRT) and Pediatric Balance Scale (PDS), and the extent to which the individual goal has been achieved will be evaluated by the Goal Attainment Scale (GAS). Assessments will be administered the day before starting treatment, after completing the 6-week Action Observation Therapy, and after a 3-month follow-up period.

Treatment Program of the Control Group (Group 1): This group will not be shown any video clips, and general physiotherapy methods will be applied to their current needs, 2 sessions a week for 6 weeks. This method includes stretching exercises for spastic muscles, strengthening exercises for the antagonist of the spastic muscle, and stabilization exercises.

Group 2: Action Observation Therapy for the lower extremities will be applied to this group by their parents at home, 2 sessions a week for 6 weeks. Participants will be shown a video of a task by their parents at home. The video to be watched will include a total of 6 activities planned to be watched every week. These 6 activities; squatting and getting up by picking up an object from the ground, walking 10 steps between parallel lines, transferring weight forward with the right and left feet, walking 5 steps sideways to the right and left, kicking the ball, climbing the step from the front and side. The video clips will be watched 3 times and after a 1-minute rest following each viewing, the participants will be asked to repeat each activity in the videos 3 times and at the end of each clip.

Group 3: Action Observation Therapy for the lower extremities will be applied by the therapist to this group, 2 sessions a week for 6 weeks. Participants will watch a video of a task presented by a therapist. The video to be watched will include a total of 6 activities planned to be watched every week. These 6 activities; squatting and getting up by picking up an object from the ground, walking 10 steps between parallel lines, transferring weight forward with the right and left feet, walking 5 steps sideways to the right and left, kicking the ball, climbing the step from the front and side. The video clips will be watched 3 times and after a 1-minute rest following each viewing, the participants will be asked to repeat each activity in the videos 3 times and at the end of each clip. After each session of Action Observation Therapy, 20 minutes of physiotherapy will be applied towards the goals of 6 activities. The scope of physiotherapy to be applied will consist of activity-based exercises for the lower extremities, stepping, weight transfer, balance and functionality.

ELIGIBILITY:
Inclusion Criteria:

- 5-13 years old

* Diagnosis of spastic hemiplegic and diplegic cerebral palsy
* Gross Motor Function Classification System (GMFCS) Level I-III
* Consent to participate in the study

Exclusion Criteria:

Exclusion criteria from the study:

* Spastic hemiplegic and diplegic disease not associated with cerebral palsy
* Presence of contractures affecting functional movement in the affected extremity
* Presence of cardiopulmonary disease or severe visual and hearing impairments
* Children who have had a seizure in the last 6 months
* Children who have had any surgery or received botulinum injections within the last 6 months or during the study period.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — men and women
Study Population: In order to prevent bias in terms of participants meeting the inclusion criteria, sociodemographic and clinical characteristics, criteria such as age, CP type, GMFCS level and presence of comorbidities were taken into account in assigning individuals to groups in the study, and the stratified randomization method will be used. Accordingly, the age ranges are taken as 5-7, 8-10, 11-13, and the CP type is; spastic diplegic and hemiplegic, GMFCS level; It will be taken as I-III and the stratification process will be done accordingly.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function measured by Gross Motor Function Measure-88 (GMFM-88) | Baseline and after 150 days
  Gross motor function will be assessed using the GMFM-88, which consists of five dimensions. The D (Standing) and E (Walking, Running, Jumping) dimensions will be used in this study. Each item is scored on a 0-3 scale, and total scores are expressed as a percentage. A higher score indicates better gross motor function. The change in GMFM-88 scores from baseline to 150 days after the intervention will be evaluated.

SECONDARY OUTCOMES:
Change in muscle tone measured by Modified Ashworth Scale (MAS) | Baseline and after 150 days
  Muscle tone will be assessed using the MAS, a 6-point ordinal scale (0-4 with 1+ as an intermediate grade) that measures resistance during passive muscle stretching in individuals with upper motor neuron lesions. A higher score indicates greater spasticity.
Change in balance function measured by Pediatric Balance Scale (PBS) | Baseline and after 150 days
  Balance function will be assessed using the PBS, which evaluates functional balance during activities requiring stability and transitions between postures. The total score ranges from 0 to 56, with higher scores indicating better balance performance.
Change in dynamic balance measured by Pediatric Reach Test (PRT) | Baseline and after 150 days
  Dynamic balance will be evaluated using the PRT, which measures the maximal reach distance in centimeters (forward, right, and left directions) while standing. Greater reach distance indicates better dynamic balance.
Change in functional mobility measured by Timed Up and Go Test (TUG) | Baseline and after 150 days
  Functional mobility will be assessed using the Timed Up and Go Test adapted for children with cerebral palsy. The time (in seconds) required to stand up from a chair, walk 3 meters, turn, return, and sit down will be recorded. A shorter time indicates better functional mobility.
Change in activity level measured by Goal Attainment Scale (GAS) | Baseline and after 150 days
  Activity levels will be assessed using the GAS, which measures achievement of individualized therapy goals. Each goal is rated on a 5-point scale from -2 (much less than expected) to +2 (much more than expected). A higher score reflects better goal attainment.
Change in participation measured by Child and Adolescent Scale of Participation (CASP) | Baseline and after 150 days
  Participation will be evaluated using the CASP, a caregiver-reported questionnaire assessing children's involvement in home, school, and community activities. The total score ranges from 0 to 100, with higher scores representing better participation.

CONTACTS AND LOCATIONS:
Overall Officials: hatice yakut, Study Director — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sgandurra G, Cecchi F, Beani E, Mannari I, Maselli M, Falotico FP, Inguaggiato E, Perazza S, Sicola E, Feys H, Klingels K, Ferrari A, Dario P, Boyd RN, Cioni G. Tele-UPCAT: study protocol of a randomised controlled trial of a home-based Tele-monitored UPper limb Children Action observation Training for participants with unilateral cerebral palsy. BMJ Open. 2018 May 14;8(5):e017819. doi: 10.1136/bmjopen-2017-017819. PMID 29764869
- [Result] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477